CLINICAL TRIAL: NCT07183449
Title: Using a Novel, User Friendly Plate Imaging System to Quantify Food Consumption in Hospitals
Brief Title: Food Quantification Using a Novel, User Friendly Plate Imaging System
Status: Recruiting | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Principal Investigator, Caroline Childs, Associate Professor, University of Southampton
Other Study IDs: IRAS Number: 343406; ERGO Number: 93184 (Other: University of Southampton)
Record Dates: First submitted 2025-09-06; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Dietary Assessment, Plate Imaging Systems, Stroke patients
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This pilot study aims to assess the feasibility of implementing a plate imaging system for dietary assessment in a stroke rehabilitation ward at University Hospital Southampton. The duration of the study is 12 weeks with an estimated sample size of 50 patients. This is a single centre study.

DETAILED DESCRIPTION:
Accurate dietary intake monitoring is essential to provide appropriate treatment for patients at risk of malnutrition, but collection of food intake data in hospital is a difficult and resource-intensive task. Paper food record charts are often incorrect or incomplete due to competing responsibilities and tasks at mealtimes, inadequate training, or removal of food trays before staff have observed intakes. Malnutrition within the hospital setting therefore continues to be under-identified and under-treated and is estimated to account for around 20% of the health and social care budget in 2023. The causes of malnutrition in hospitals are multifactorial and include acute illness or disease, dislike of food, and psychosocial or environmental factors. Approaches trialled in clinical settings to optimise dietary intakes of patients to date include protected mealtimes, dedicated mealtime assistance, and changes to the presentation and preparation of food. Across the literature, poor food intake and malnutrition was highly correlated with poor patient outcomes. In line with the NHS long-term plan and the UHS digital team's plan for a paperless digital Trust, a digital dietary assessment tool would provide a valid and reliable tool to accurately monitor dietary intakes. Electronic records will enable examination of longitudinal changes in intakes and/or dietary quality, and to identify patterns of intakes associated with positive or negative clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who eat hospital food
* Patients with a capacity to give consent
* Non-English-speaking patients with interpreters
* Patients who are aged 18 years and above

Exclusion Criteria:

* Patients who receive exclusive parenteral or enteral nutrition
* Patients who do not eat hospital provided meals
* Patients on end-of-life care plan
* Patients who do not give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to the stroke rehabilitation ward will be proposed to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional Intake | Week 1 up to week 12 of the study
  Nutritional intake in calories (kcal), macronutrients and micronutrients as measured by the plate imaging system

SECONDARY OUTCOMES:
Length of stay | From week 1 up to week 12 of study
  Length of stay in hospital as measured by the date of admission to the ward to the date of discharge from the ward.
Weight | From week 1 up to week 12 of the study
  Weight as measured on the date of admission to the ward to the date of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Caroline E Childs, BSc (Hons), PhD, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardenas D, Bermudez C, Perez A, Diaz G, Cortes LY, Contreras CP, Pinzon-Espitia OL, Gomez G, Gonzalez MC, Fantin R, Gutierrez J, Sulz I, Tarantino S, Hiesmayr M. Are traditional screening tools adequate for monitoring the nutrition risk of in-hospital patients? An analysis of the nutritionDay database. JPEN J Parenter Enteral Nutr. 2022 Jan;46(1):83-92. doi: 10.1002/jpen.2085. Epub 2021 Mar 10. PMID 33554364
- [Background] Trtovac D, Lee J. The Use of Technology in Identifying Hospital Malnutrition: Scoping Review. JMIR Med Inform. 2018 Jan 19;6(1):e4. doi: 10.2196/medinform.7601. PMID 29351894
- [Background] Young AM, Banks MD, Mudge AM. Improving nutrition care and intake for older hospital patients through system-level dietary and mealtime interventions. Clin Nutr ESPEN. 2018 Apr;24:140-147. doi: 10.1016/j.clnesp.2017.12.009. Epub 2018 Jan 3. PMID 29576353
- [Background] Future Health. (2023). Hiding in plain sight: Tackling malnutrition as part of the prevention agenda. Available at Hiding-in-plain-sight-Web-FINAL-Nov-2023.pdf (futurehealth-research.com)
- [Background] Heelan, A. R. (2021). A mixed methods study to determine the feasibility of providing finger foods for patients after stroke in hospital. University of Southampton, Doctoral Thesis, 330pp. https://eprints.soton.ac.uk/484431/
- [Background] Thibault R, Abbasoglu O, Ioannou E, Meija L, Ottens-Oussoren K, Pichard C, Rothenberg E, Rubin D, Siljamaki-Ojansuu U, Vaillant MF, Bischoff SC. ESPEN guideline on hospital nutrition. Clin Nutr. 2021 Dec;40(12):5684-5709. doi: 10.1016/j.clnu.2021.09.039. Epub 2021 Oct 20. PMID 34742138